CLINICAL TRIAL: NCT02419729
Title: Evaluation of Fractional CO2 Laser Treatment Efficacy and Comparison to Vaginal Estrogen Therapy in Postmenopausal Women With Vulvovaginal Atrophy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Faculdade de Medicina do ABC (Other)
Responsible Party: Principal Investigator, Vera Lucia, Principal Investigator, Faculdade de Medicina do ABC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 39495014.0.0000.0082
Record Dates: First submitted 2015-04-06; First posted 2015-04-17 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Vulvovaginal Atrophy
Keywords: Vulvovaginal atrophy; Menopause; Fractional CO2 laser; Estrogen cream
MeSH Terms: interventions — Lasers, Gas; Estrogens; Estriol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- CO2 laser & Estrogen (Experimental): Effective fractional CO2 laser therapy and effective estrogen vaginal cream
  Interventions: Device: CO2 laser; Drug: Estrogen
- CO2 laser & Placebo of Estrogen (Active Comparator): Effective fractional CO2 laser therapy and placebo of estrogen vaginal cream.
  Interventions: Device: CO2 laser; Drug: Placebo of Estrogen
- Placebo of CO2 laser & Estrogen (Sham Comparator): Placebo fractional CO2 laser therapy and effective estrogen vaginal cream.
  Interventions: Drug: Estrogen; Device: Placebo of CO2 laser

INTERVENTIONS:
Device: CO2 laser — SMARTXIDE2 V2LR (DEKA-Pulse) was used in each application using minimal parameters suggested by the laser's software ( Power of 30 W, 1000us emission time, 1000um spacing and a level of SmartStack 2)
  Other Names: Fractionated CO2 laser
  Arms: CO2 laser & Estrogen; CO2 laser & Placebo of Estrogen
Drug: Estrogen — Topical estrogen cream treatment: Estriol 1mg daily.
  Other Names: Estriol 1mg
  Arms: CO2 laser & Estrogen; Placebo of CO2 laser & Estrogen
Drug: Placebo of Estrogen — Placebo of topical estrogen cream.
  Arms: CO2 laser & Placebo of Estrogen
Device: Placebo of CO2 laser — SMARTXIDE2 V2LR (DEKA-Pulse) was used in each applications using minimal parameters suggested by the laser's software but power of 0.5 W was stipulated for the placebo intervention and other parameters remained unchanged.
  Other Names: SMARTXIDE2 V2LR - Monalisa Touch - Deka Laser
  Arms: Placebo of CO2 laser & Estrogen

SUMMARY:
Forty-five women will be included in a double-blind randomized trial in order to compare fractional CO2 laser treatment, local estrogen therapy and the combination of both treatments for Vulvovaginal Atrophy (VVA) and determine the efficacy and possible adverse effects CO2 laser treatment.

DETAILED DESCRIPTION:
Vulvovaginal atrophy (VVA) symptoms are strongly associated with declining ovarian function and estrogen levels in postmenopausal women, having a considerable impact on women's life quality. Topical hormonal therapy and hormonal replacement are widely used to alleviate VVA symptoms. In this context, minimal invasive fractional CO2 laser emerges as an alternative non-hormonal therapy, especially in patients that present contraindications to hormonal therapy. Objective: Compare fractional CO2 laser treatment, local estrogen therapy and the combination of both treatments for VVA and determine the efficacy and possible adverse effects CO2 laser treatment. Materials and Methods: Forty-five postmenopausal women will be randomized in three double-blinded groups of treatment consisting of CO2 laser and placebo of estrogen vaginal cream, placebo of CO2 laser and estrogen vaginal cream and CO2 laser and estrogen vaginal cream. Assessment of baseline characteristics and follow-up will be obtained through self-completion questionnaires (Female Sex Function Index, International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF), Vulvovaginal Symptom Questionnaire and The Menopause-Specific Quality of Life (MENQOL)). Frost Index and Vaginal Health Index (VHI) are part of objective clinical and histologic analyses. Colposcopy, vaginal cytology and middle third lateral vaginal wall biopsy will also be performed at baseline and at week 17.

ELIGIBILITY:
Inclusion Criteria:

* 45-65 women with amenorrhea for over 24 months.
* Clinical vaginal atrophy diagnosis.

Exclusion Criteria:

* BMI > 35.
* Previous use of oral estrogen therapy in the last 6 months.
* History or current diagnosis of cancer.
* Altered cervical smear in the last 12 months.
* Renal or hepatic insufficiency.
* Drug-induced menopause.
* Previous use of steroids.
* Previous vaginal radiotherapy therapy.
* Vulvovaginitis.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-03; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Vulvovaginal Symptom Questionnaire | Baseline, week 10 and week 17
  Vulvovaginal Symptom Questionnaire will be used to evaluate improvement of vulvovaginal atrophy symptoms.

SECONDARY OUTCOMES:
Vaginal Cytology Improvement | Baseline, week 10 and week 17
  Vaginal cytology will be obtained from the middle third lateral vaginal wall in order to evaluate initial conditions of the vaginal wall and modifications after treatment. Frost Index, Karyopyknotic Index and Eosinophilic Index will be applied to each sample to measure improvement of vaginal atrophy.
Change from Baseline in Female Sex Function Index | Baseline, week 10 and week 17
  Female Sex Function Index will be used to evaluate improvement of vulvovaginal atrophy symptoms.
Change from Baseline in The Menopause-Specific Quality of Life | Baseline, week 10 and week 17
  The Menopause-Specific Quality of Life will be used to evaluate improvement of vulvovaginal atrophy symptoms.

OTHER OUTCOMES:
Urinary Incontinence Improvement | Baseline, week 10 and week 17
  Incontinence Questionnaire-Short Form (ICIQ-SF) will be used in order to evaluate urinary incontinence improvement after treatment.
Vaginal Health Index Improvement | Baseline, week 10 and week 17
  Evaluation of vaginal wall conditions such as pH, elasticity, bleeding signs, secretion type and consistency and hydration.

CONTACTS AND LOCATIONS:
Overall Officials: Vera L da Cruz, MD, Principal Investigator — Faculdade de Medicina do ABC
Locations (1):
- Centro de Atencao a Saude da Mulher, São Bernardo do Campo, São Paulo, Brazil

REFERENCES:
- [Result] Salvatore S, Nappi RE, Parma M, Chionna R, Lagona F, Zerbinati N, Ferrero S, Origoni M, Candiani M, Leone Roberti Maggiore U. Sexual function after fractional microablative CO(2) laser in women with vulvovaginal atrophy. Climacteric. 2015 Apr;18(2):219-25. doi: 10.3109/13697137.2014.975197. Epub 2014 Dec 16. PMID 25333211
- [Result] Society of Obstetricians and Gynaecologists of Canada. SOGC clinical practice guidelines. The detection and management of vaginal atrophy. Number 145, May 2004. Int J Gynaecol Obstet. 2005 Feb;88(2):222-8. doi: 10.1016/j.ijgo.2004.11.003. PMID 15779109
- [Result] Bachman GA. A new option for managing urogenital atrophy in post-menopausal women. Cont Obstet Gynecol 42, pp. 13-28.
- [Result] Salvatore S, Nappi RE, Zerbinati N, Calligaro A, Ferrero S, Origoni M, Candiani M, Leone Roberti Maggiore U. A 12-week treatment with fractional CO2 laser for vulvovaginal atrophy: a pilot study. Climacteric. 2014 Aug;17(4):363-9. doi: 10.3109/13697137.2014.899347. Epub 2014 Jun 5. PMID 24605832
- [Derived] Ippolito GM, Crescenze IM, Sitto H, Palanjian RR, Raza D, Barboglio Romo P, Wallace SA, Orozco Leal G, Clemens JQ, Dahm P, Gupta P. Vaginal lasers for treating stress urinary incontinence in women. Cochrane Database Syst Rev. 2025 Jul 25;7(7):CD013643. doi: 10.1002/14651858.CD013643.pub2. PMID 40709601